CLINICAL TRIAL: NCT06424795
Title: Molecular and Microbiome/Metagenome Correlates of Recurrent Wheeze in RSV Infected Infants
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Mary Caserta, Professor of Pediatrics, University of Rochester
Other Study IDs: MISP 58711-062022-002
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Syncytial Virus Infection
Keywords: wheeze
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two anterior nasal swabs and a nasal brush. Samples retained only if agreed to by Legally Authorized Representative on Parent Permission form
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants with recurrent wheeze: Infants with recurrent wheeze in the year following primary RSV infection
- Infants without recurrent wheeze: Infants without recurrent wheeze in the year following primary RSV infection

SUMMARY:
The goal of this observational study is to learn about further wheezing in infants with RSV infection.. The main question it aims to answer is:

If infant factors, the infant immune response in the nose and the bacteria that reside in the nose at the time of primary RSV infection can predict/classify infants with recurrent wheezing during the following year.

A secondary aim is to identify infant immune response factors in the nose and patterns of bacteria in the nose during primary RSV infection that may help us understand why recurrent wheezing occurs.

Researchers will compare infants with repeated episodes of wheezing to infants who do not have further wheezing.

Participants will be full term infants with their first RSV infection. We will collect information on the pregnancy and birth history as well as the signs and symptoms of RSV infection. Two nasal swabs and a nasal wash will be collected from the infants. Six weeks following the RSV infection we will begin contact with the families biweekly to determine if the infant has recurrent wheezing confirmed by a medical provider. Follow-up will continue for approximately 1 year, through a second winter season.

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) causes yearly epidemics of respiratory infection with a significant burden of disease in those at the extremes of age. Infants with RSV infection develop a range of illness from mild or in apparent upper respiratory infections to severe lower respiratory disease with wheezing and/or pneumonia. RSV infection is the most common cause of hospitalization in infants in the US.

The great majority (85%) of hospitalized infants are diagnosed with bronchiolitis and 78% are noted to have wheezing. RSV infection leads to even greater outpatient utilization of medical care including Emergency Department visits (39-69 per 1000 under 6 months and 45-68 per 1000 from 6-11 months) and visits to pediatricians (108-157/1000 under 6 months and 160-194 per 1000 from 6-11 months).

Following primary RSV infection several epidemiological observations have identified an increased frequency of recurrent wheezing in 34 to 56% of infants.

The objectives of this study include:

Primary Objective: To test whether clinical factors, airway gene expression and microbiome/metagenome patterns in the nasal epithelium at the time of primary RSV infection can predict/classify infants with recurrent wheezing.

Secondary Objective 1: To identify airway gene expression and microbiome/metagenome correlates of primary RSV infection that may inform pathogenic mechanisms associated with recurrent wheeze.

Hypotheses

Primary Hypothesis: Infants with recurrent wheeze following primary RSV infection will have a defined set of clinical, airway gene expression and/or airway microbiome/metagenome characteristics associated with a post bronchial wheezing phenotype.

Secondary Hypothesis 1: Respiratory epithelial innate immune responses to primary RSV infection, and their interaction with microbiome composition and functional processes, will identify biological mechanisms contributing to post bronchial wheeze.

This is a single center, prospective, case-control observational study. Full term (>36 and 0/7 gestation) infants born after the prior RSV season of the prior year with primary RSV infection and no prior episodes of wheezing will be enrolled during their first RSV season from both outpatient and inpatient locations in Rochester New York. During the subsequent seasons of enrollment infants will meet the above eligibility requirements and also be tested and negative for acute infection with Severe Acute Respiratory Syndrome-Coronavirus-2.100 infants total with RSV infection will be enrolled with approximately 50 from the hospital and 50 from the Emergency Department (ED) or outpatient clinic in order to enroll infants with a range of severity, but with a focus on those presenting for medical care due to symptoms. Active surveillance for subsequent wheezing episodes will be conducted by phone/text/email follow-up every two weeks over the subsequent year, including a second full winter season for all subjects, beginning six weeks after the index illness. At the first report of subsequent wheezing a research clinic or home visit will be conducted to confirm the presence of wheezing by a trained staff member. Recurrent wheeze will be defined by two separate episodes of wheezing separated by at least 14 days with the first episode confirmed by study staff. In addition to this active surveillance, caregiver's will be asked to sign a medical records release for their child at the first visit that will cover the period of participation in the study. At the end of the study we will review each subject's medical records to determine if the child has had wheezing documented by a medical provider and not reported by the family. Once recurrent wheeze has been confirmed the subject will have reached an endpoint. At the end of the follow-up period the clinical and biological characteristics of participants with recurrent wheeze and those without recurrent wheeze will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by Legally Authorized Representative
2. Confirmed infection with RSV
3. Gestational age at birth 36 and 0/7 weeks or greater
4. No prior wheezing episodes
5. Negative for acute infection with SARS-CoV-2
6. First RSV season

Exclusion Criteria:

1. Underlying disease (immune, cardiopulmonary, neuromuscular, renal) that would qualify for palivizumab
2. Receiving immunosuppressive medications
3. Live greater than 35 miles from University of Rochester Medical Center
4. Parental inability to read or understand English

Ages: 3 Days to 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will enroll previously healthy infants born after 36 0/7 weeks gestation during their first RSV infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-12-21 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Medically confirmed recurrent wheeze | Follow-up for recurrent wheeze begins 6 weeks after the primary RSV infection and ends approximately one year later (including a subsequent RSv season).
  Recurrent wheezing documented by a medical provider following primary RSV infection

CONTACTS AND LOCATIONS:
Overall Officials: Mary T Caserta, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hall CB, Weinberg GA, Iwane MK, Blumkin AK, Edwards KM, Staat MA, Auinger P, Griffin MR, Poehling KA, Erdman D, Grijalva CG, Zhu Y, Szilagyi P. The burden of respiratory syncytial virus infection in young children. N Engl J Med. 2009 Feb 5;360(6):588-98. doi: 10.1056/NEJMoa0804877. PMID 19196675
- [Background] Turi KN, Shankar J, Anderson LJ, Rajan D, Gaston K, Gebretsadik T, Das SR, Stone C, Larkin EK, Rosas-Salazar C, Brunwasser SM, Moore ML, Peebles RS Jr, Hartert TV. Infant Viral Respiratory Infection Nasal Immune-Response Patterns and Their Association with Subsequent Childhood Recurrent Wheeze. Am J Respir Crit Care Med. 2018 Oct 15;198(8):1064-1073. doi: 10.1164/rccm.201711-2348OC. PMID 29733679